CLINICAL TRIAL: NCT00345696
Title: Phase II Study of First Line Capecitabine Administered on Continuous Way Combined With Oxaliplatin and Bevacizumab Every Two Weeks in Metastatic Colorectal Cancer Patients.
Brief Title: 1stline Study Capecitabine Administered on Continuous Way Plus Oxaliplatin&Bevacizumab Every 2weeks in Metastatic CCR.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unidad Integral de Investigación en Oncología S.L. (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XELOXAVBISEMANAL
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Capecitabine; Oxaliplatin; Bevacizumab; First line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/Kg intravenous, 90-60-30 minutes, every 2 weeks.
  Other Names: Avastin
Drug: Capecitabine — 600 mg/m2, orally, every 12 hours, continuous.
  Other Names: Xeloda
Drug: Oxaliplatine — 85 mg/m2, intravenous, 2 hours infusion, every 2 weeks
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to determinate progression free survival after 9 months of treatment.

DETAILED DESCRIPTION:
To look for a new chemotherapy management to get less acute and chronic toxicity and/or an easier administration treatment line.

This study tries to demonstrate an alternative chemotherapy scheme,continuous polychemotherapy regimen with less dose with the added effect of the monoclonal antibody Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > or = 18 years
* Outpatients with ECOG performance status ≤ 2.
* Histologically confirmed diagnosis of CRC patients with metastasis.
* Presence of at least one detectable lesion in accordance with RECIST criteria.
* Life expectancy greater than 3 months.
* Patients who are able to understand the study request and want to participate.
* Written informed consent given

Exclusion Criteria:

* Patients who have been treated with Bevacizumab previously.
* Received any systemic treatment previously to treat an advanced or metastatic disease
* Adjuvant or neoadjuvant treatment to non-metastatic disease is allowed, provided that there has been finished at least 6 months before the initial study treatment.
* If the patient has been treated with adjuvant therapy previously, it is not allowed to be included in the study in case of disease progression during the treatment or during 6 months later than the end of the treatment.
* If radiotherapy has been administered it has not been administered in the lesion selected for the study, and the end of the treatment has been finished at least 4 weeks before the study initiation.
* Previous surgical procedure of the IV stage disease is allowed.
* PAst or current history (within the last 5 years) of malignancies except curatively treated basal and squamous cell carcinoma of the skin, and in-situ carcinoma of the cervix.
* History or evidence upon physical examination of central nervous system (CNS) (i.e. primary cerebral tumour, uncontrolled convulsions with standard medical treatment, cerebral metastasis or any kind or ictus history).
* History of psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant cardiovascular disease (active), i.e, uncontrolled hypertension, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication or peripheral vascular disease. Patients have undergone myocardial infarction in the previous year of the study initiation will be excluded.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to take oral medications
* Patients subjected to allogenic transplant and request immunotherapy.
* Bone fracture not healed, wounds or severe ulcers.
* Known hemorrhagic diathesis or coagulopathy.
* Uncontrolled and severe intercurrent infections or another severe and uncontrolled concomitant diseases.
* Moderate or severe renal impairment (creatinine clearance < 30 ml/min (calculated according to Cockroft-Gault formula) or serum creatinine >1,5 x ULN.
* Any of the following laboratory values:

Absolute neutrophils count (ANC) < 1.5 x 109/l. Platelet count < 100 x 109/l. Hemoglobin < 9 g/dl. INR > 1.5. Total bilirubin > 1.5 ULN. ALT and/or AST > 2.5 x ULN or > 5 x ULN (in case of hepatic metastasis). Alkaline phosphatase > 2.5 x ULN or >5 x ULN (in case of hepatic metastasis), or > 10 x ULN (in case of bone metastasis).

* History of unexpected serious adverse events to fluoropyrimidine treatments or known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patients subjected to major surgical procedure, open biopsy or who had significant traumatic injures in 28 days time before the start of the study treatment , or patients with a major surgery procedure planning during the study period. Fine needle aspiration biopsy 7 days before the study initiation.
* Use of full dose of oral or parenteral anticoagulants ( at least 10 days before the start of the study treatment or thrombolytic agents. Low dose of warfarin is allowed, with an INR ≤ 1.5.
* Subject requiring chronic use of high dose aspirin (> 325 m/day) or non-steroidal anti-inflammatory treatment.
* Participation in another treatment trial within 4 weeks of the study initiation.
* Pregnant (serum positive pregnancy test) or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 9 months

SECONDARY OUTCOMES:
Overall Response rate | 24 months
Overall survival | 24 months
Toxicity of the combination of capecitabine+oxaliplatin+bevacizumab | 24 months
Resection rate of hepatic or pulmonary metastases | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Grávalos, MD, Study Chair — Unidad Integral de Investigación en Oncología S.L.; Cristina Grávalos, MD, Principal Investigator — Hospital 12 de Octubre
Locations (1):
- Hospital 12 de Octubre, Madrid, Madrid, Spain